CLINICAL TRIAL: NCT06530875
Title: The Effect of Training on Childhood Vaccines Given to Expectant Mothers on Vaccine Hesitation and Vaccine Literacy: A Randomised Controlled Experimental Study
Brief Title: Vaccination Hesitation in Expectant Mothers
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, Eda Nur MUHAFİZ, NURSE, Yuzuncu Yil University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Yüksek Lisans Tez
Record Dates: First submitted 2024-07-28; First posted 2024-07-31 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Vaccine Hesitation
Keywords: Vaccine Hesitancy; Vaccine Literacy; Immunization; Child; Pediatric Nursing
MeSH Terms: conditions — Vaccination Hesitancy

STUDY DESIGN:
Intervention Model Description: The research was planned as a cross section (pre-test post-test, experimental and control group) randomized controlled study.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arms (Experimental): The experimental group will be trained on hesitations in childhood vaccines.
  Interventions: Behavioral: training on hesitations regarding childhood vaccinations
- Control (No Intervention): there will be no interference

INTERVENTIONS:
Behavioral: training on hesitations regarding childhood vaccinations — Training will be given to expectant mothers on childhood vaccination hesitations
  Arms: Arms

SUMMARY:
The aim of this study is to increase the awareness of vaccination with the training on childhood vaccine hesitancy given to expectant mothers by a nurse during pregnancy. In addition, it is aimed to evaluate the effect of the training given to expectant mothers on vaccine hesitancy and vaccine literacy.

Hypotheses of the study

H0: Training on Childhood Vaccine Hesitancy does not affect vaccine hesitancy and vaccine literacy in expectant mothers.

H1a: Education on Childhood Vaccine Hesitancy affects vaccine hesitancy in expectant mothers.

H1b: Education on Childhood Vaccine Hesitancy affects vaccine literacy in expectant mothers.

DETAILED DESCRIPTION:
Vaccination, which is one of the basic elements of preventive health services, is the most effective, safe and cost-effective health practice in protecting human health and preventing infectious diseases. Vaccination has been recognized as the most effective method for people to cope with infectious diseases. Vaccines protect infants and children against many diseases. Every year, 1 million 700 thousand people die in the world due to vaccine-preventable diseases (Odabaş & Kuzlu Ayyıldız, 2021).

Despite scientific and historical evidence of the safety and effectiveness of vaccines and immunization, some groups are still hesitant and reluctant to accept vaccines and immunization. The concept of vaccine hesitancy was defined by the World Health Organization Strategic Advisory Group of Experts on Immunization (SAGE) Vaccine Hesitancy Working Group: "vaccine hesitancy is recognized as the delay or refusal to accept vaccines despite the availability of immunization services". These behaviors include refusal, delay or reluctant acceptance despite active concerns (Etesaminia & Derinpınar, 2021). In our country, since 2010, negative media news about vaccines started to affect families and "vaccine refusal" started to be observed. As of 2015, the rates of vaccine refusal started to increase with the winning of the lawsuit on "obtaining parental consent for vaccine administration". While 183 families refused vaccination in 2011, 980 families in 2013, 5,400 families in 2015, 12,000 families in 2016 and 23,000 families in 2018 refused to vaccinate their children. It is stated that if the number of families refusing vaccines reaches 50 thousand, childhood infectious diseases that have been reduced or eradicated may cause an epidemic (Çıtak & Aksoy, 2020). In this context, scientific studies should be conducted on the effects and side effects of vaccines, and effective communication and trust between parents and health personnel will be one of the most effective ways to eliminate hesitations about vaccination. In addition, the use of mass media and social media in informing and raising public awareness about the results of scientific studies on vaccines and their effects will enable rapid progress in the fight against "anti-vaccination". It is suggested that health personnel should be informed and raised awareness about the subject in order to make parents more aware of vaccine administration, appropriate vaccine counseling services should be provided for families against those who make anti-vaccine discourses, and educational programs can be prepared to increase the level of knowledge of parents about vaccines. (Argın et al., 2022).

Vaccine literacy encompasses the knowledge, motivation and competence to access, understand, evaluate and apply health information in order to make the right health decisions in daily life. Individuals with adequate vaccine literacy accept vaccination as a sine qua non of a functioning health system, undertake the task of vaccine advocacy in every environment they are in, and develop an uncomplicated system to ensure vaccine communication with other people (Şahin & Baran Aksakal, 2022).

In a study, most of the participants stated that they obtained information about vaccines from the internet. Mothers emphasized that they frequently used social media for vaccines and other health issues, and that they were concerned about the information accessed and doubted about vaccines (Çıklar & Döner, 2020). In a study examining the relationship between parents' e-health literacy and confidence in vaccines, it was found that parents' confidence in vaccines decreased as the e-health literacy level increased (Ceylan et al., 2022), while in another study examining the relationship between parents' health literacy and their attitudes and behaviors towards childhood vaccines, it was found that parents' health literacy level was not related to their attitudes and behaviors towards childhood vaccines (Ertuğrul & Albayrak, 2021). In another study conducted with university students, it was found that as the health literacy level of university students increased, their anti-vaccine attitudes decreased (Ertaş & Göde, 2021).

In a study, it was stated that the rate of vaccine refusal has reached serious dimensions, that this rate will increase further if measures are not taken, and that the most important of these measures is education. Therefore, it was reported that it is important to organize trainings on vaccines, especially in family health centers that provide primary health care services, and that active use of the media by health personnel on vaccination and vaccination is also required. at the same time, it was suggested that these trainings can also be done by meeting face to face with parents. as a result, it was reported that parents will be made aware of vaccination and a decrease in the rate of vaccine refusal will be observed (Huseynov, 2021).

The aim of this study is to increase the awareness of vaccination with the training on childhood vaccine hesitancy given to expectant mothers by a nurse during pregnancy. In addition, it is aimed to evaluate the effect of the training given to expectant mothers on vaccine hesitancy and vaccine literacy.

ELIGIBILITY:
Inclusion Criteria:

* Pregnancy over 18 years of age
* Literacy
* Volunteering to participate in the study

Exclusion Criteria:

* Adolescent pregnancy (under 18 years of age)
* Communication problems
* Having any psychiatric problem
* Having a chronic disease
* illiteracy
* Not volunteering to participate in the study

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Vaccine Literacy Scale for Childhood Vaccines | 3 weeks
  The Vaccine Literacy Scale consists of 3 sub-dimensions and 13 items in total: Functional Health Literacy, Communicative Health Literacy and Critical Health Literacy.

SECONDARY OUTCOMES:
Vaccine Hesitation Scale | 3 weeks
  The vaccine hesitancy scale consists of 10 items. Items 1, 2, 3, 4, 6, 7 and 8 contain positive statements, while items 5, 9 and 10 contain negative statements. While the level of vaccine hesitancy decreases as the degrees given by the participants to the positive statements increase, the level of vaccine hesitancy increases as the degrees given to the negative statements increase.

CONTACTS AND LOCATIONS:
Overall Officials: Yuzuncu Y University, Study Director — Yuzuncu Yil University
Locations (1):
- Yuzuncu Yıl University, Van, Turkey (Türkiye)